CLINICAL TRIAL: NCT00564252
Title: The Efficacy of Topical Finasteride in the Treatment of Idiopathic Hirsutism
Brief Title: Topical Finasteride in the Treatment of Idiopathic Hirsutism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Collaborators: Firuzgar hospital affiliated to Iran University of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 84-5-6886; IUMS127
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Idiopathic Hirsutism
MeSH Terms: interventions — Finasteride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: topical finasteride — 0.2%topical(cream)finasteride twice a day for six months

SUMMARY:
the purpose of this study is to evaluate the efficacy of topical Finasteride in the treatment of idiopathic hirsutism

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic hirsutism which is defined as normal levels of androgens and normal ovulation
* Normal serum prolactin

Exclusion Criteria:

* Pregnancy
* Simultaneous use of other drugs for the treatment of hirsutism

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-02; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
the efficacy of topical finasteride was determined by comparison of Ferriman-Gallwey score before and after medication | 6 months

SECONDARY OUTCOMES:
the efficacy of topical finasteride was determined by comparison of mean hair thickness before and after medication | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: iraj heydari, professor assistant, Study Director — endocrine and metabolism centre of Iran University of Medical Sciences